CLINICAL TRIAL: NCT02604407
Title: A Phase 3, Randomized, Double-blind, Multicenter, Placebo-controlled, Forced-dose Titration, Safety and Efficacy Study of SHP465 in Adults Aged 18-55 Years With Attention-deficit/ Hyperactivity Disorder (ADHD)
Brief Title: Safety and Efficacy Study of SHP465 in Adults Aged 18-55 Years With Attention-deficit/ Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHP465-306
Record Dates: First submitted 2015-11-11; First posted 2015-11-13 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- SHP465 12.5 mg (Experimental): Subjects will receive SHP465 12.5 mg
  Interventions: Drug: SHP465 12.5mg capsules (one capsule daily)
- SHP465 37.5 mg (Experimental): Subjects will receive SHP465 titrated up to 37.5 mg
  Interventions: Drug: SHP465 12.5mg, 25mg, or 37.5mg capsules (one capsule daily)
- Placebo (Placebo Comparator): Subjects will receive matching placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SHP465 12.5mg capsules (one capsule daily) — one capsule daily
  Arms: SHP465 12.5 mg
Other: Placebo — Matching placebo capsule that appears identical in size, weight, shape, and color (one capsule daily)
  Arms: Placebo
Drug: SHP465 12.5mg, 25mg, or 37.5mg capsules (one capsule daily) — One capsule daily
  Arms: SHP465 37.5 mg

SUMMARY:
The study is designed to evaluate the efficacy and safety of each dose of SHP465 (12.5 and 37.5 mg) given to participants daily in the morning compared to placebo in the treatment of adults aged 18 to 55 years diagnosed with ADHD.

ELIGIBILITY:
Inclusion Criteria:

Subject must be 18-55 years of age

Subject is able to provide written, personally signed and dated informed consent.

Subject is willing and able to comply with all of the testing and requirements defined in the protocol

Subject, who is a female, must not be pregnant.

Subject must have a satisfactory medical assessment with no clinically significant or relevant abnormalities.

Subject has a primary diagnosis of ADHD.

Subject has an adult ADHD-RS with prompts total score ≥28 at the baseline visit.

Subject must have a minimum level of intellectual functioning, as determined by the investigator.

Subject is able to swallow a capsule.

Subject is currently not on ADHD therapy or is not completely satisfied with any aspect of their current ADHD therapy.

Exclusion Criteria:

Subject has a current, comorbid psychiatric diagnosis with significant symptoms.

Subject is considered a suicide risk in the opinion of the investigator

Subject has a body mass index (BMI) of <18.5 kg/m2 at the screening visit.

Subject has a BMI ≥40 kg/m2 at the screening visit.

Subject has a concurrent chronic or acute illness, disability, or other condition.

Subject has a history of seizure, a chronic or current tic disorder, or a current diagnosis of Tourette's disorder.

Subject has a history of moderate to severe hypertension.

Subject has a known history of symptomatic cardiovascular disease

Subject has a known family history of sudden cardiac death or ventricular arrhythmia.

Subject has any clinically significant ECG or clinically significant laboratory abnormality at the screening visit.

Subject has current abnormal thyroid function

Subject has a documented allergy, hypersensitivity, or intolerance to amphetamine or to any excipients in the investigational product.

Subject has failed to respond, to an adequate course(s) of amphetamine therapy.

Subject has a history of suspected substance abuse or dependence disorder.

Subject has a positive urine drug result at the screening visit (with the exception of subject's current stimulant therapy, if any) or Subject has taken another investigational product or has taken part in a clinical study within 30 days prior to the screening visit.

Subject has previously completed, has discontinued, or was withdrawn from this study.

Subject is taking any medication that is excluded or has not been appropriately washed out according to the protocol requirements.

Subject is required to take or anticipates the need to take medications that have CNS effects or affect performance.

Subject is female and is pregnant or lactating.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 275 (Actual)
Dates: Start 2015-11-19 (Actual); Primary Completion 2016-03-24 (Actual); Study Completion 2016-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (45):
- United States (45):
  - Pharmacology Research Institute, Encino, California
  - Pharmacology Research Institute (Pri), Los Alamitos, California
  - Pharmacology Research Institute (Pri), Newport Beach, California
  - Nrc Research Institute, Orange, California
  - Elite Clinical Trials, Wildomar, California
  - McB Clinical Research, Colorado Springs, Colorado
  - Florida Clinical Research Center Llc, Bradenton, Florida
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Clinical Neuroscience Solutions, Inc, Jacksonville, Florida
  - Florida Clinical Research Center, Llc, Maitland, Florida
  - Qps Mra, Llc, Miami, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Clinical Neuroscience Solutions, Inc, Orlando, Florida
  - Northwest Behavioral Research Center, Marietta, Georgia
  - Capstone Clinical, Libertyville, Illinois
  - Baber Research Group, Inc, Naperville, Illinois
  - Psychiatric Associates, Overland Park, Kansas
  - Louisiana Research Associates, Inc., New Orleans, Louisiana
  - Rochester Center For Behavioral Medicine, Rochester Hills, Michigan
  - Clinical Neurophysiology Services, Sterling Heights, Michigan
  - Psychiatric Care and Research Center, O'Fallon, Missouri
  - Midwest Research Group, Saint Charles, Missouri
  - Premier Psychiatric Research Institutute, Lincoln, Nebraska
  - Center For Psychiatry and Behavioral Medicine, Inc, Las Vegas, Nevada
  - Princeton Medical Institute, Princeton, New Jersey
  - Bioscience Research Llc, Mount Kisco, New York
  - Nyu Langone Medical Center, New York, New York
  - Richard H Weisler, Md, Pa & Associates, Raleigh, North Carolina
  - Midwest Clinical Research Center, Dayton, Ohio
  - Ips Research Company, Oklahoma City, Oklahoma
  - Oregon Center For Clinical Investigations, Inc, Portland, Oregon
  - Oregon Center For Clinical Investigations, Salem, Oregon
  - Omega Medical Research, Warwick, Rhode Island
  - Rainbow Research, Inc., Barnwell, South Carolina
  - Coastal Carolina Research, Mt. Pleasant, South Carolina
  - Clinical Neuroscience Solutions, Memphis, Tennessee
  - Futuresearch Trials of Dallas, Lp, Dallas, Texas
  - Bayou City Research, Ltd, Houston, Texas
  - Red Oak Psychiatry Associates, Houston, Texas
  - Houston Clinical Trials, Llc, Houston, Texas
  - Research Across America, Plano, Texas
  - Neuroscience, Inc, Herndon, Virginia
  - Eastside Therapeutic Resource, Kirkland, Washington
  - Summit Research Network (Seattle) Llc, Seattle, Washington

REFERENCES:
- [Derived] Weisler RH, Greenbaum M, Arnold V, Yu M, Yan B, Jaffee M, Robertson B. Efficacy and Safety of SHP465 Mixed Amphetamine Salts in the Treatment of Attention-Deficit/Hyperactivity Disorder in Adults: Results of a Randomized, Double-Blind, Placebo-Controlled, Forced-Dose Clinical Study. CNS Drugs. 2017 Aug;31(8):685-697. doi: 10.1007/s40263-017-0455-7. PMID 28712074

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 43 study centers in the United States between 19 November 2015 and 24 March 2016.
Pre-assignment Details: A total of 369 participants were screened and 275 participants were enrolled in the study.
Groups:
- Placebo: Participants received placebo matched to SHP465 capsule orally once daily for 4 weeks.
- SHP465 12.5 mg: Participants received SHP465 capsule 12.5 milligram (mg) orally once daily for 4 weeks.
- SHP465 37.5 mg: Participants received SHP465 capsule of 12.5 mg during week 1 and 25 mg at week 2 followed by 37.5 mg at weeks 3 and 4 orally once daily.
Period: Overall Study
Arm/Group | Placebo | SHP465 12.5 mg | SHP465 37.5 mg
Started | 91 | 92 | 92
TREATED | 89 | 92 | 90
Completed | 80 | 80 | 76
Not Completed | 11 | 12 | 16
Not completed — Adverse Event | 0 | 7 | 5
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 5
Not completed — Lost to Follow-up | 2 | 1 | 2
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Other | 3 | 1 | 4

BASELINE CHARACTERISTICS:
Population: Safety set consisted of all participants in the randomized set (participants who signed informed consent for whom a randomization number had been assigned) who had taken at least 1 dose of investigational product.
Groups:
- SHP465 12.5 mg: Participants received SHP465 capsule 12.5 mg orally once daily for 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | SHP465 12.5 mg | SHP465 37.5 mg | Total
Number analyzed (Participants) | 89 | 92 | 90 | 271
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.5 (10.77) | 33 (10.40) | 32.4 (10.02) | 33.3 (10.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 35 | 39 | 121
  Male | 42 | 57 | 51 | 150

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Adult Attention-deficit/Hyperactivity Disorder Rating Scale-4 (ADHD-RS) With Prompts Total Score at Visit 6 (Week 4)
Description: The ADHD-RS was developed to measure the behaviors of children with Attention deficit hyperactivity disorder (ADHD). The adult ADHD-RS with prompts consists of 18 items designated to reflect current symptomatology of ADHD based on the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria. Each item is scored on a 4-point scale ranging from 0 (no symptoms) to 3 (severe symptoms), with the total score for the rating scale ranging from 0 to 54. Higher score = more severe symptoms.The scale is subdivided into 2 subscales of 9 symptoms each: hyperactivity/impulsivity and inattentiveness. Adult prompts are included with the ADHD-RS to create a semistructured measurement that allows the clinician to probe the extent, frequency, breadth, severity, and consequences of these symptoms to ascertain impairment in an adult population.
Time Frame: Baseline, Visit 6 (Week 4)
Population: Full Analysis Set (FAS) consisted of all participants in the safety set who had at least 1 post dose baseline primary efficacy assessment (ADHD-RS with prompt total score) on treatment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | SHP465 12.5 mg | SHP465 37.5 mg
Number analyzed (Participants) | 86 | 89 | 88
Units on a scale
  Baseline | 40.5 (6.52) | 39.8 (6.38) | 39.9 (7.07)
  Change at Visit 6: number analyzed (Participants) | 77 | 78 | 73
  Change at Visit 6 | -11.0 (11.47) | -18.1 (13.42) | -23.8 (11.89)
Statistical Analysis 1: Comparison: Placebo vs SHP465 12.5 mg; Test type: Superiority or Other; p < 0.001, Mixed-effects model for repeated measure; Difference of LS Mean = -8.1, 95% CI 2-sided [-11.7 to -4.4] — Between treatment groups of SHP465 12.5 mg and Placebo
Statistical Analysis 2: Comparison: Placebo vs SHP465 37.5 mg; Test type: Superiority or Other; p < 0.001, Mixed-effects model for repeated measure; Difference of LS Mean = -13.4, 95% CI 2-sided [-17.1 to -9.7] — Between treatment groups of SHP465 37.5 mg and Placebo

2. Secondary Outcome: Clinical Global Impression of Improvement (CGI-I) Score at Visit 6 (Week 4)
Description: CGI scales permit a global evaluation of the participant's severity and improvement over time. CGI-I was performed to rate the severity of a participant's condition on a 7-point scale ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill participants).
Time Frame: Visit 6 (Week 4)
Population: Full-analysis set (FAS) consisted of all participants in the safety set who had at least 1 postdose baseline primary efficacy assessment (ADHD-RS with prompt total score) on treatment with number of participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | SHP465 12.5 mg | SHP465 37.5 mg
Number analyzed (Participants) | 77 | 78 | 73
Units on a scale | 3.1 (1.05) | 2.4 (1.16) | 1.9 (1.10)

ADVERSE EVENTS:
Time Frame: From the Start of Study Drug Administration up to Follow-up (Week 5)
Arm/Group | Placebo | SHP465 12.5 mg | SHP465 37.5 mg
Serious Adverse Events (participants affected / at risk) | 0/89 | 0/92 | 0/90
Other Adverse Events (participants affected / at risk) | 12/89 | 44/92 | 49/90
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=89) | SHP465 12.5 mg (N=92) | SHP465 37.5 mg (N=90)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 13 (13) | 20 (20)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 18 (18) | 27 (27)
Headache (Nervous system disorders) | 4 (4) | 6 (6) | 11 (11)
Anxiety (Psychiatric disorders) | 1 (1) | 6 (7) | 4 (4)
Bruxism (Psychiatric disorders) | 0 (0) | 1 (1) | 5 (5)
Initial insomnia (Psychiatric disorders) | 1 (1) | 4 (4) | 6 (6)
Insomnia (Psychiatric disorders) | 1 (1) | 12 (12) | 10 (13)
Irritability (Psychiatric disorders) | 0 (0) | 5 (6) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.